CLINICAL TRIAL: NCT06410157
Title: Cardiac-Control Affecting Learning Through Mindfulness (CALM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Irvine (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mara Mather, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP-21-00357-main; R01AG080652 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Age-related Cognitive Decline; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increase Oscillation (Experimental): Participants will breath at a slow "resonance" frequency during a breath-focused mindfulness practice and receive biofeedback to increase heart rate oscillation.
  Interventions: Behavioral: Daily practice
- Decrease Oscillation (Experimental): Participants' breathing will not be fixed to particular frequency during a breath-focused mindfulness practice and they will receive biofeedback to decrease heart rate oscillation.
  Interventions: Behavioral: Daily practice

INTERVENTIONS:
Behavioral: Daily practice — Participants will be asked to undergo daily mindfulness practice while regulating (either increase or decrease) heart rate oscillation.

SUMMARY:
Some types of meditation lead heart rate to become more steady as breathing quiets whereas others lead to large heart rate swings up and down (oscillations) as breathing becomes deeper and slower. The current study is designed to investigate how daily mindfulness practice with heart rate biofeedback during breathing in a pattern that either increases or decreases heart rate oscillation affect attention and memory and blood biomarkers associated with Alzheimer's disease.

ELIGIBILITY:
Inclusion criteria

* Fluent in English
* Black/African-American or White/European-American
* Aged between 50-70 years old
* Non-pregnant and non-menstruating (for at least the past year)
* Have normal or corrected-to-normal vision and hearing
* Have reliable access to wifi
* Have an email account that you check regularly
* Have a phone that receives text messages
* Agree to provide blood and urine samples at two campus visits
* Agree to devote up to 50 minutes daily to this study for 10 weeks as well as attend two campus visits

Exclusion criteria

* Have a disorder that would impede performing the breathing intervention (e.g., abnormal cardiac rhythm, arrhythmia, dyspnea)
* Have cognitive impairment
* Have regularly played Lumosity games in the past 6 months
* Have any conditions listed below that are not safe for MRI

  * *Metal in any parts of your body
  * Claustrophobia
  * Have worked as a machinist, metal worker, or in any profession or hobby grinding metal?
  * Have had an injury to the eye involving a metallic object (e.g., metallic slivers, shavings, or foreign body)
  * Cardiac pacemaker
  * Implanted cardiac defibrillator
  * Aneurysm clip or brain clip
  * Carotid artery vascular clamp
  * Neurostimulator
  * Insulin or infusion pump
  * Spinal fusion stimulator
  * Cochlear, otologic, ear tubes or ear implant
  * Prosthesis (eye/orbital, penile, etc.)
  * Implant held in place by a magnet
  * Heart valve prosthesis
  * Artificial limb or joint
  * Other implants in body or head
  * Electrodes (on body, head or brain)
  * Intravascular stents, filters
  * Shunt (spinal or intraventricular)
  * Vascular access port or catheters
  * IUD
  * Transdermal delivery system or other types of foil patches (e.g., Nitro, Nicotine, Birth control, etc.) that cannot be removed for MRI
  * Shrapnel, buckshot, or bullets
  * Tattooed eyeliner or eyebrows
  * Body piercing(s) that cannot be removed for MRI
  * Metal fragments (eye, head, ear, skin)
  * Internal pacing wires
  * Aortic clips
  * Metal or wire mesh implants
  * Wire sutures or surgical staples
  * Harrington rods (spine)
  * Bone/joint pin, screw, nail, wire, plate
  * Wig or toupee that cannot be removed for MRI
  * Hair implants that involve staples or metal
  * Hearing aid(s) that cannot be removed for MRI
  * Dentures or retainers that cannot be removed for MRI

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in plasma amyloid-beta 42 levels | Week 1 and Week 10
  Plasma Ab42 levels will be compared for Week 1 (pre-intervention) and Week 10 (post-intervention). Investigators will test for a time X condition interaction in plasma Ab 42 levels (to assess group differences in change).

SECONDARY OUTCOMES:
Plasma amyloid-beta 40 levels | Week 1 and Week 10
  Plasma Ab40 levels will be compared for Week 1 (pre-intervention) and Week 10 (post-intervention). Investigators will test for a time X condition interaction in plasma Ab 40 levels (to assess group differences in change).
Plasma Ab42/40 ratio | Week 1 and Week 10
  Investigators will test for a time X condition interaction with plasma Ab42/40 ratio values as the dependent variable (to assess group differences in change).
Plasma pTau-181/tTau ratio | Week 1 and Week 10
  Investigators will test for a time X condition interaction with the ratio of pTau-181 and total tau values as the dependent variable (to assess group differences in change).
Change in brain perivascular space volume | Week 1 and Week 10
  Investigators will test for a time X condition interaction in perivascular space volume.
Brain training performance on Lumosity games during the breathing intervention | During intervention (daily during Weeks 2-10) and before intervention (daily during Week 1)
  Investigators will compute a general learning factor across performance on all games played daily during the intervention period (Weeks 2-10) and separately across performance on all games played daily before the intervention period (Week 1). Investigators will test for group differences in performance during the intervention, controlling for performance before the intervention.

OTHER OUTCOMES:
Locus coeruleus (LC) responses to novel faces | Week 1 and Week 10
  Investigators will test for a time x condition interaction in phasic LC responses to novel faces during an fMRI face-name task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual scores associated with the primary and secondary outcomes will be shared.
  Functional and structural brain images will be shared. Lumosity game play data will be shared.
Time Frame: IPD will be shared upon publication of results from those IPD with no end date.
Access Criteria: The investigators plan to use Openneuro.org, but if options change, the investigators may select another database. The plan is to have the data shared at a repository where those who are interested can access it. At Openneuro.org, all data are freely available to all users.